CLINICAL TRIAL: NCT07099287
Title: TRANSformá tu Salud Dejando de Fumar: Advancing Smoking Cessation Among Transgender
Brief Title: Advancing Smoking Cessation Among Transgender
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Fundación Huésped (Other)
Responsible Party: Principal Investigator, Francisco Cartujano, MD, Assistant Professor - Department of Public Health Sciences (SMD), University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FH-077; R21CA284313 (NIH)
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRANSform your health (Experimental): A culturally adapted smoking cessation intervention for transgender and gender diverse individuals living in Argentina
  Interventions: Behavioral: TRANSform your health

INTERVENTIONS:
Behavioral: TRANSform your health — A culturally adapted smoking cessation intervention for transgender and gender diverse individuals living in Argentina

SUMMARY:
In partnership with a Community Advisory Board, the investigators developed TRANSformá tu salud (Spanish for TRANSform your health), a culturally adapted smoking cessation intervention for transgender and gender diverse individuals living in Argentina. This was a single-arm pilot study with 40 TGD individuals who smoke and received TRANSformá tu salud. The investigators assessed the feasibility, acceptability, and preliminary impact of TRANSformá tu salud.

DETAILED DESCRIPTION:
In partnership with a Community Advisory Board, the investigators developed TRANSformá tu salud (Spanish for TRANSform your health), a culturally adapted smoking cessation intervention for transgender and gender diverse individuals living in Argentina. This was a single-arm pilot study with 40 TGD individuals who smoke and received TRANSformá tu salud. The investigators assessed the feasibility, acceptability, and preliminary impact of TRANSformá tu salud.

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals self-identified as transgender and gender diverse individuals, were 18 years old or older, smoked at least three days per week, were interested in quitting smoking within the next 30 days, had an active cellphone with WhatsApp®, and were willing to complete two study visits.

Exclusion Criteria:

* Use of other tobacco products (including e-cigarettes), pregnancy or breast-feeding, plans to move from their current residence in the next six months, and shared residence with a current study participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Transgender and gender diverse individuals
Enrollment: 40 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-02-05 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Reporting 7-Day Point Prevalence Smoking Abstinence at Month 3 | Month 3
  Seven-day point prevalence smoking abstinence is defined as no cigarette smoking, not even a puff, during the 7 days prior to the Month 3 assessment. Abstinence will be assessed as a binary outcome (yes or no), and the result will be reported as the percentage of participants who meet this criterion at Month 3.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Cartujano, MD, Principal Investigator — University of Rochester
Locations (1):
- Fundación Huésped, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No